CLINICAL TRIAL: NCT07071337
Title: A Randomized, Open-label, Multicenter Phase III Clinical Study of SKB264 Versus Investigator's Choice of Chemotherapy in Subjects With Unresectable Locally Advanced, Relapsed, or Metastatic Hormone Receptor-positive (HR+)/Human Epidermal Growth Factor Receptor 2-negative (HER2-) Breast Cancer Who Have Previously Failed Endocrine Therapy
Brief Title: A Study of SKB264 Versus Investigator's Choice of Chemotherapy in Subjects With Unresectable Locally Advanced, Relapsed, or Metastatic HR+/HER2- Breast Cancer Who Have Previously Failed Endocrine Therapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-Ⅲ-13
Record Dates: First submitted 2025-06-19; First posted 2025-07-17 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer
Keywords: SKB264; HR+/HER2- breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Paclitaxel; Capecitabine

STUDY DESIGN:
Intervention Model Description: Participants will be randomised in a 1:1 ratio to one of two intervention groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SKB264 (Experimental)
  Interventions: Drug: SKB264
- Investigator's Choice of Chemotherapy (Active Comparator): Nab-paclitaxel, paclitaxel or capecitabine will be administered and managed according to the investigator's clinical judgment, guided by clinical practice.
  Interventions: Drug: Nab-paclitaxel; Drug: Paclitaxel; Drug: Capecitabine

INTERVENTIONS:
Drug: SKB264 — 5mg/kg, IV on Day 1 and Day 15 of each 28 day cycle
  Arms: SKB264
Drug: Nab-paclitaxel — 100 mg/m^2, IV, on Days 1, 8, and 15 every 4 weeks
  Arms: Investigator's Choice of Chemotherapy
Drug: Paclitaxel — 90 mg/m^2, IV, on Days 1, 8, and 15 every 4 weeks; or 80 mg/m^2, IV, weekly, every 3 weeks
  Arms: Investigator's Choice of Chemotherapy
Drug: Capecitabine — 1000-1250 mg/m^2, orally, Days 1-14, twice daily, every 3 weeks
  Arms: Investigator's Choice of Chemotherapy

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SKB264 in patients with unresectable locally advanced, recurrent, or metastatic HR+/HER2- breast cancer who have previously failed endocrine therapy.

DETAILED DESCRIPTION:
This is a randomized, open-label, multicenter phase 3 clinical study to evaluate the efficacy and safety of SKB264 monotherapy versus investigator's choice of chemotherapy (ICC) in subjects with unresectable locally advanced, recurrent, or metastatic HR+/HER2- breast cancer who had failed at least one line of systemic chemotherapy and have not recieved systemic chemotherapy for locally advanced, relapsed, or metastatic stages.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥ 18 and ≤ 75 years at the time of signing the ICF, male or female;
2. Histologically and/or cytologically confirmed HR+/HER2- BC based on pathological reports from the most recent biopsy or other pathological specimens;
3. Subjects must have radiologically documented disease progression during or after the most recent treatment prior to enrollment;
4. No prior systemic chemotherapy for locally advanced, relapsed, or metastatic stages. Subjects who previously received adjuvant/neoadjuvant chemotherapy and progressed >6 months after completion of the last chemotherapy treatment will be allowed for study inclusion;
5. The investigator assessed that the patient could not continue to benefit from endocrine therapy and was suitable for receiving first-line chemotherapy;
6. Able to provide recently newly obtained or archival tumor tissue sections at or after diagnosis of relapsed or metastatic tumor within the recent prior to randomization;
7. At least one measurable lesion per RECIST v1.1；
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 with no worsening within 2 weeks prior to randomization;
9. Life expectancy of ≥ 12 weeks;
10. Suitable to receive one of the chemotherapy regimens listed in the investigator's choice of chemotherapy (paclitaxel, nab-paclitaxel, capecitabine) as assessed by the investigator;
11. Adequate organ and bone marrow function;
12. Having recovered from all toxicities due to prior treatment;
13. Use of effective medical contraception during study treatment and for 6 months after the end of dosing for female subjects of childbearing potential and male subjects with partners of childbearing potential;
14. Willingness to participate in the study, sign the ICF, and comply with the protocol-specified visits and relevant procedures.

Exclusion Criteria:

1. Subjects with locally advanced breast cancer suitable for curative therapy at study enrollment;
2. Other malignancies (except those tumors cured by local treatment, such as basal cell carcinoma of skin, squamous cell carcinoma of skin, carcinoma in situ of the cervix) within 3 years prior to randomization;
3. Subiects with known meningeal metastases, brainstem metastases, spinal cord metastases and/or compression or active centralnervous system (CNS) metastases.
4. Presence of any serious cardiovascular and cerebrovascular diseases or cardiovascular and cerebrovascular risk factors;
5. History of (noninfectious) interstitial lung disease (ILD)/noninfectious pneumonitis requiring steroid therapy and current ILD/noninfectious pneumonitis, or suspected ILD/noninfectious pneumonitis at screening that cannot be excluded by imaging;
6. Clinically serious lung injuries caused by lung diseases;
7. Serious infection within 4 weeks prior to randomization, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia; active infection requiring systemic anti-infective therapy within 2 weeks prior to randomization;
8. Documented severe dry eye syndrome, severe meibomian gland dysfunction and/or blepharitis, or history of severe corneal disorders that prevent/delay corneal healing;
9. History of esophagogastric varices, severe ulcers, gastric perforation, gastrointestinal obstruction, intra-abdominal abscess, or acute gastrointestinal bleeding within 6 months prior to randomization;
10. Active hepatitis B (hepatitis B surface antigen positive and HBV-DNA ≥ 500 IU/mL or above the ULN, whichever is higher) or hepatitis C (hepatitis C antibody positive and HCV-RNA above the ULN);
11. Positive result of human immunodeficiency virus (HIV) test or history of acquired immunodeficiency syndrome (AIDS); known active syphilis infection;
12. 12 Known hypersensitivity to SKB264 or investigator's choice chemotherapy or any of its excipients, including but not limited to polysorbate-20, or history of severe hypersensitivity reaction to other monoclonal antibodies;
13. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
14. Pregnant or lactating women;
15. Prior TROP2-targeted therapy or any treatment containing chemotherapeutic agents targeting topoisomerase I (including antibody-drug conjugates [ADCs]);
16. Live vaccines within 4 weeks prior to randomization or scheduled to receive live vaccines during study treatment;
17. Receipt of the following therapies prior to randomization: a)Major surgery within 4 weeks prior or expected major surgery during the study; b)Radiation therapy within 2 weeks prior (extensive radiation therapy including radiopharmaceuticals within 4 weeks prior); c)Any immunotherapy, biological therapy, or other investigational drugs within 4 weeks or 5 half-lives of prior drug use (whichever is shorter) (bisphosphonates or RANK-L inhibitors for bone metastases are permitted prior to randomization); or traditional Chinese medicine with approved anti-tumor indications, small molecule targeted therapy, or endocrine therapy within 2 weeks prior.
18. Rapid deterioration of the condition, e.g., significant changes in performance status, etc., during the screening process.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2025-07-18 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) assessed by Blinded Independent Central Review (BICR) | Randomization up to approximately 24 months
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on BICR or death due to any cause, whichever occurs first

SECONDARY OUTCOMES:
Overall Survival (OS) | Randomization up to approximately 67 months
  OS is defined as the time from randomization until the date of death due to any cause
Progression-Free Survival (PFS) assessed by Investigator | Randomization up to approximately 24 months
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on investigator or death due to any cause, whichever occurs first.
Objective Response Rate (ORR) | Randomization up to approximately 24 months
  ORR is defined as the percentage of patients who achieve complete response(CR) or partial response (PR), as assessed by BICR/investigator per RECIST 1.1
Disease control rate (DCR) | Randomization up to approximately 24 months
  DCR is defined as the percentage of patients who achieve CR, PR or stable disease (SD), as assessed by BICR/ investigator per RECIST 1.1
Duration of Response (DoR) | Randomization up to approximately 24 months
  DoR is defined as the time from the date of first documented CR or PR until date of documented disease progression per RECIST 1.1, as assessed by BICR/investigator or death due to any cause, whichever occurs first.
Time to Response (TTR) | Randomization up to approximately 24 months
  TTR is defined as the time from the date of randomization until the first documentation of CR or PR as assessed by BICR/investigator per RECIST 1.1.
AEs and SAEs | AEs should be collected from signing the informed consent form (ICF) until 30 days after the last dose
  Incidence and severity of AEs and SAEs (per CTCAE 5.0), and clinically significant abnormal laboratory findings
Mean change from baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Randomization up to approximately 24 months
  To assess the impact of SKB264 on disease related symptoms and health related quality of life (HRQoL) in this patient population
Mean change from baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Breast Cancer Module 23 (EORTC QLQ-BR23) | Randomization up to approximately 24 months
  To assess the impact of SKB264 on disease related symptoms and health related quality of life (HRQoL) in this patient population
Anti-drug Antibodies (ADA) for SKB264 | Day1 and Day15 of Cycle 1 (each cycle is 28 days), Day1 of Cycle 3, Cycle 6, and so on (every 3 cycles), up to approximately 24 months
  Immunogenicity test results and titer values of SKB264
Maximum observed plasma concentration (Cmax) of SKB264-ADC, SKB264-TAB and free KL610023 | Day1 and Day15 of Cycle 1 (each cycle is 28 days), Day1 of Cycle 3, Cycle 6, and so on (every 3 cycles), up to approximately 24 months
  To assess the pharmacokinetic (PK) profile of SKB264.
Minimum observed plasma concentration (Cmin) of SKB264-ADC, SKB264-TAB and free KL610023 | Day1 and Day15 of Cycle 1 (each cycle is 28 days), Day1 of Cycle 3, Cycle 6, and so on (every 3 cycles), up to approximately 24 months
  To assess the pharmacokinetic (PK) profile of SKB264.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Fifth Medical Center of the Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong